CLINICAL TRIAL: NCT02510001
Title: A Sequential Phase I Study of MEK1/2 Inhibitors PD-0325901 or Binimetinib Combined With cMET Inhibitor PF-02341066 in Patients With RAS Mutant and RAS Wild Type (With Aberrant c-MET) Colorectal Cancer
Brief Title: MEK and MET Inhibition in Colorectal Cancer
Acronym: MErCuRIC1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Queen's University, Belfast (Other); Oxford University Hospitals NHS Trust (Other); Velindre NHS Trust (Other Government); University Hospital, Antwerp (Other); Hospital Vall d'Hebron (Other); Saint Antoine University Hospital (Other); European Georges Pompidou Hospital (Other); Pfizer (Industry); University of Turin, Italy (Other); Belfast Health and Social Care Trust (Other); Beaumont Hospital (Other); European Commission (Other); Array BioPharma (Industry); University of Paris 5 - Rene Descartes (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OCTO-049
Record Dates: First submitted 2015-06-18; First posted 2015-07-28 (Estimated); Results first posted 2021-04-26 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-01

CONDITIONS: Solid Tumor; Colorectal Cancer
Keywords: RASMT CRC; RASWT/c-MET CRC; Dose Escalation; Histologically or cytologically confirmed; Dose Expansion
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Crizotinib; mirdametinib; binimetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- Dose Escalation Phase Cohort 1 Dose level 1 (Experimental): Crizotinib 250mg OD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day1, then Day 1-21 every 28 day cycle
  Interventions: Drug: PF-02341066; Drug: PD-0325901
- Dose Escalation Phase Cohort 2 Dose level 2 (Experimental): Crizotinib 200mg BD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day1, then Day 1-21 every 28 day cycle
  Interventions: Drug: PF-02341066; Drug: PD-0325901
- Dose Escalation Phase Cohort 3 Dose level 3 (Experimental): Crizotinib 200mg BD Days 1-28 continuously PD-0325901 4mg BD Run in Day -7 to Cycle 1 Day 1, then Day 1-21 every 28 day cycle
  Interventions: Drug: PF-02341066; Drug: PD-0325901
- Dose Escalation Phase Cohort 4 Dose level 4 (Experimental): Crizotinib 200mg BD Days 1-28 continuously PD-0325901 8mg BD Run in Day -7 to Cycle 1 Day1, then Day 1-21 every 28 day cycle
  Interventions: Drug: PF-02341066; Drug: PD-0325901
- Dose Escalation Phase Cohort 7 Dose level 5 (Experimental): Binimetinib 30mg BD continuous administration or Days 1-21 every 28 days. PF-02341066 200mg BD continuous administration
  Interventions: Drug: PF-02341066; Drug: PD-0325901; Drug: Binimetinib
- Dose Escalation Phase Cohort 13 Dose level 5a (Experimental): Binimetinib 30mg BD interval dose administration Days 1-21 every 28 days. PF-02341066 250mg OD continuous administration
  Interventions: Drug: PF-02341066; Drug: Binimetinib
- Dose Expansion Phase (Experimental): Binimetinib 30mg BD interval dose administration Days 1-21 every 28 days PF-02341066 (Crizotinib) 250mg OD Days 1-28 continuously Dosage determined following the recommended Phase II dose identification in the dose escalation phase.
  Interventions: Drug: PF-02341066; Drug: Binimetinib
- Dose Escalation Phase Cohort 12 Dose level 5 (Interval dosing) (Experimental): Binimetinib 30mg BD interval dose administration days 1-21 every 28 days. PF-02341066 200mg BD continuous administration
  Interventions: Drug: PF-02341066; Drug: Binimetinib

INTERVENTIONS:
Drug: PF-02341066 — PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  Other Names: Crizotinib
Drug: PD-0325901 — PD-0325901 2mg - 8mg BD with Run in Day -7 to Day-1 on Cycle 1 Day1, then Day 1-21 every 28 day cycle.
  Other Names: No other Intervention name for this drug
  Arms: Dose Escalation Phase Cohort 1 Dose level 1; Dose Escalation Phase Cohort 2 Dose level 2; Dose Escalation Phase Cohort 3 Dose level 3; Dose Escalation Phase Cohort 4 Dose level 4; Dose Escalation Phase Cohort 7 Dose level 5
Drug: Binimetinib — Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
  Other Names: MEK162
  Arms: Dose Escalation Phase Cohort 12 Dose level 5 (Interval dosing); Dose Escalation Phase Cohort 13 Dose level 5a; Dose Escalation Phase Cohort 7 Dose level 5; Dose Expansion Phase

SUMMARY:
This trial is designed to try two new cancer drugs together for the first time. The investigators think that they might be effective in some types of bowel cancer. The first part of the trial will see what doses of the two drugs can safely be given together. Once the investigators have identified a suitable dose combination they will look at how effective treatment is in bowel cancers where either the RAS gene is mutated, or MET is over-active. In the trial the investigators will look at samples of blood, skin and tumour to check the drugs are working in the way expected. The trial will take place in three sites in the UK and 5 sites in Europe. The trial is funded as part of the European commission's FP7 program.

DETAILED DESCRIPTION:
This is a two stage study. Firstly a dose escalation step is used to define the best dose for the drug combination, using the rolling 6 design where up to 6 patients are recruited at each dose level, and increasing the dose of one or other agent according to the side effects of treatment. An initial dose escalation phase was completed where 25 patients were enrolled, using the study treatment combination of PD-0325901 with PF-02341066. Following discontinuation of the MEKi (inihibitor), PD-0325901, the study was updated to include a further dose escalation phase using the new combination study treatment, MEKi, Binimetinib with METi, PF-02341066. The effects of this drug combination will be assessed to define the recommended dose level for the dose expansion phase of the study.

Second the new drug combination is observed in 42-98 patients with bowel cancer for its efficacy and tolerability. Patients who give consent will have their archival tumour samples tested for RAS and c-MET status.

Potential participants will, after giving consent, undergo screening tests to ensure that it is safe for them to take part. These involve a detailed medical history, physical exam, blood tests, ophthalmology exam, ECG and ultrasound and skin biopsies. The size and extent of tumours is also assessed by CT and/or MRI scan.

For the initial dose escalation phase, on assurance that the test results are satisfactory, patients start on PD-0325901 first for one week. On Day -7 a physical exam, ECG and blood test is performed, with a repeat blood test on Day -6. End of first week PD samples of blood are taken to observe the level of PD-0325901. Day 1 PF-02341066 is introduced after further clinical safety assessments. There are further blood samples taken over 24 hours to measure levels of PD-0325901 and PF-02341066 on days 21 and 28 of the first cycle.

For the further dose escalation phase, again assuming that the screening test results are satisfactory, patients start on Day 1 with the combined treatment of PF-02341066 with Binimetinib. A physical exam, ECG and blood test is performed, with a repeat blood test on Day 2. There are further blood samples taken over 24 hours to measure levels of Binimetinib and PF-02341066 on day 21of the first cycle.

Patients have weekly visits when side effects are reviewed and a physical examination is performed. On Day 15 a second skin biopsy is taken along with blood tests to assess liver and renal function. At the end of the first 4 weeks cycle, for the initial dose escalation phase, and at end of 8 weeks for the new combination therapy dose escalation phase, an ophthalmology exam is compared with the baseline assessment.

For subsequent cycles in both the initial dose escalation and further dose escalation phases, visits remain weekly and include safety assessments as per Day 1. Blood levels of PD-0325901 or Binimetinib and PF-02341066 are measured on day 21 of even numbered cycles. In addition the tumour size is checked every second cycle, and the study treatment stopped if the tumour continues to grow.

When patients stop taking the study treatment they will be reviewed after 4 weeks for any side effects and have a physical examination and other safety tests performed.

For patients entering the expansion phase of the trial the procedures are similar, except that there is a pre-screening stage where tumour biopsies are required. Patients will have a sample of their tumour assessed, following consent, to determine their RAS and cMET status. This may involve a fresh biopsy. If suitable, the patient will be entered into the screening for the dose expansion phase and a fresh tumour biopsy may be taken if not already done so. The study schedule is the same as for the escalation phase using Binimetinib with PF-02341066. At the end of treatment a further, optional, tumour biopsy may be taken.

After trial participation patients will be offered further care with the trial team or their referring oncology team as appropriate.

ELIGIBILITY:
INCLUSION CRITERIA (Inclusion criteria for the completed initial dose escalation phase using PF-02341066/PD-0325901 are listed in Appendix 7.) All patients

* Age ≥ 16 years (>18 years in France)
* ECOG performance status 0-1 (Appendix 1)
* Adequate respiratory function on clinical assessment
* Left ventricular ejection fraction (LVEF) ≥ 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram┼
* Able to give informed consent prior to any screening procedures being performed and be capable of complying with the protocol and its requirements
* Haematological and biochemical indices within the ranges shown below:
* Haemoglobin (Hb) ≥ 9g/dl (transfusion to achieve this allowed ),
* Neutrophils ≥ 1,500/μl,
* Platelet count ≥ 100,000/μl,
* AST or ALT ≤ 2.5 x ULN, patient with liver metastases ≤ 5 × ULN,
* Alkaline phosphatase ≤ 5 x ULN,
* Serum Bilirubin ≤ 1.5 x ULN,
* Creatinine Clearance ≥ 50ml/min (Calculated by Cockcroft Gault equation, or by EDTA) (Appendix 2)
* Able to swallow oral medication
* Life expectancy of at least 3 months.

Dose escalation phase:

* Patients with any advanced solid tumours
* Patients for whom the combination of PF-02341066 with Binimetinib is a reasonable option.

Dose expansion phase:

Patients will be eligible for pre-screening for this phase provided that:

* They have given informed consent to screening.
* They are willing to undergo a biopsy for assessment of tumour RAS mutation status and c-MET assessment.
* The Investigator anticipates that they are likely to satisfy the eligibility criteria for the trial. Formal screening should not be performed until the tumour pre-screening result is known.

Eligibility for the trial, in patients passing pre-screening, requires:

* Histologically confirmed colorectal adenocarcinoma that is either a) RASMT (KRAS codon 12, 13, 61, 117, 146; NRAS codon 12, 13, 61, 117, 146) or b) RASWT/c-MET mutated/amplified or c) RASWT/c-MET over-expressed with progressive disease on or within 6 months of completion of adjuvant therapy or after chemotherapy and/or targeted therapies for metastatic disease.
* Prior treatment with an EGFR targeted monoclonal antibody for patients with RASWT/c-MET mutated or amplified CRC or c) RASWT/c-MET over-expressed CRC.
* No evidence for a mutation in BRAF at codon600
* Metastases accessible for biopsy on 2-3 occasions
* At least one other measurable lesion (according to RECIST v1.1).
* Unsuitable for potential curative resection. ┼For non-UK territories: if echocardiogram (ECHO) cannot be performed, a MUGA scan may be performed in compliance with local policy, applicable national legislation and relevant approvals. Cardiac ejection fraction must be determined as measured by ECHO in the UK.

EXCLUSION CRITERIA (Exclusion criteria for the completed initial dose escalation phase using PF-02341066/PD-0325901 are listed in Appendix 7.) All patients

* Unstable ischaemic heart disease, cardiac dysrhythmias, coronary/peripheral artery bypass graft or cerebrovascular accident within 6 months prior to starting treatment.
* Uncontrolled arterial hypertension despite medical treatment.
* Ongoing congestive heart failure or cardiac dysrhythmias of NCI CTCAE Grade ≥2 or uncontrolled atrial fibrillation.
* History of extensive disseminated/bilateral or known presence of Grade 3 or 4 interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, interstitial lung disease (ILD), obliterative bronchiolitis, and pulmonary fibrosis. A history of prior radiation pneumonitis is allowed.
* Any active central nervous system (CNS) lesion (i.e., those with radiographically unstable, symptomatic lesions) and/or leptomeningeal metastases. However, patients treated with stereotactic radiotherapy or surgery are eligible if the patient remained without evidence of CNS disease progression ≥ 3 months. Patients must be off corticosteroid therapy for ≥ 3 weeks.
* Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy);
* Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. NB: Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on Binimetinib treatment
* Spinal cord compression unless treated with the patient attaining good pain control and stable or recovered neurologic function.
* Carcinomatous meningitis or leptomeningeal disease.
* History of hypoalbuminaemia, or patients with peritoneal disease or pleural disease, where there is a requirement for ascitic or pleural taps.
* History of retinal vein occlusion, intraocular pressure > 21 mmHg or patient considered at risk of retinal vein thrombosis (e.g. history of hyperviscosity or hypercoagulability syndromes).
* History of retinal degenerative disease.
* History of Gilbert's syndrome.
* Active infections (including chronic hepatitis type B or C and HIV infection if status known), severe immunologic defect, compromised bone marrow function.
* Other severe acute or chronic medical (including severe gastro-intestinal disorders e.g. partial bowel obstruction, malabsorption, active inflammatory bowel disease) or psychiatric conditions or laboratory abnormalities that the investigator considers would make the patient a poor trial candidate, would impart excess risk associated with study participation or drug administration or could interfere with protocol compliance or the interpretation of trial results.
* Patients who have undergone major surgery ≤ 3 weeks prior to starting study drug or who have not recovered from side effects of such procedure.
* Use of drugs or foods that are known potent CYP3A4 inhibitors or inhibitors or are CYP3A4 substrates with narrow therapeutic indices (see Appendix 5).
* Radiotherapy (except for palliative reasons), endocrine therapy, immunotherapy or chemotherapy during the previous four weeks (six weeks for nitrosoureas, Mitomycin-C) and four weeks for investigational medicinal products before treatment. Patients with prostate cancer may continue to receive endocrine therapy to maintain castrate levels of androgens.
* Resting ECG with QTc > 480msec at 2 or more time points within a 24h period (using Fredericia correction).
* Requirement for medication known to prolong QT interval (Appendix 5).
* History of other malignancy less than 3 years before the diagnosis of current cancer, EXCLUDING the following: Non-melanoma skin cancer, in situ carcinoma of the cervix treated surgically with curative intent, other malignant tumours that have been treated curatively and patient is deemed disease-free
* Women with the ability to become pregnant (or already pregnant or lactating). However, those female patients who have a negative serum pregnancy test before enrolment and agree to use one highly effective form of contraception (oral, injected or implanted hormonal contraception or intra-uterine device) in addition to condom plus spermicide for four weeks before entering the trial, during the trial and for six months afterwards are considered eligible.
* Male patients with partners of child-bearing potential unless they agree to take measures not to father children by using one form of highly effective contraception including oral, injected or implanted hormonal contraception or intra-uterine device in addition to condom plus spermicide, during the trial and for six months afterwards). Men with pregnant or lactating partners should be advised to use barrier method contraception (condom plus spermicidal gel) to prevent exposure to the foetus or neonate.
* Prior exposure to any of a HGF, cMET or a MEK inhibitor.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-12-03 (Actual); Study Completion 2018-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Middleton, Principal Investigator — Oxford University Hospital NHS Trust
Locations (1):
- Oxford University Hospital NHS Trust, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about the trial on the Oncology Clinical Trials Office (OCTO) website. — http://www.oncology.ox.ac.uk/trial/mercuric1

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 patient in escalation phase dose 5 was registered to the trial on 28Sep2016 but withdrew before dose administration due to unexpected and fast disease progression.
Groups:
- Dose Escalation Phase Dose 1.: Crizotinib (PF-02341066) 250mg OD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day -1, then Day 1-21 every 28 day cycle
- Dose Escalation Phase Dose 2.: Crizotinib (PF-02341066) 200mg BD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day -1, then Day 1-21 every 28 day cycle
- Dose Escalation Phase Dose 3.: Crizotinib (PF-02341066) 200mg BD Days 1-28 continuously PD-0325901 4mg BD Run in Day -7 to Cycle 1 Day 1, then Day 1-21 every 28 day cycle
- Dose Escalation Phase Dose 4.: Crizotinib (PF-02341066) 200mg BD Days 1-28 continuously PD-0325901 8mg BD Run in Day -7 to Cycle 1 Day -1, then Day 1-21 every 28 day cycle
- Dose Escalation Phase 5.: Binimetinib 30mg BD continuous administration or Days 1-21 every 28 days. Crizotinib (PF-02341066) 200mg BD continuous administration
- Dose Escalation Phase Dose 5a: Binimetinib 30mg BD interval dose administration Days 1-21 every 28 days. Crizotinib (PF-02341066) 250mg OD continuous administration
- Dose Escalation Phase Dose 5 (Interval Dosing): Binimetinib 30mg BD interval dose administration days 1-21 every 28 days. Crizotinib (PF-02341066) 200mg BD continuous administration
Period: Overall Study
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4. | Dose Escalation Phase 5. | Dose Escalation Phase Dose 5a | Dose Escalation Phase Dose 5 (Interval Dosing) | Dose Expansion Phase
Started | 6 | 5 | 6 | 8 | 8 | 7 | 5 | 37
Completed | 6 | 5 | 6 | 6 | 4 | 5 | 3 | 30
Not Completed | 0 | 0 | 0 | 2 | 4 | 2 | 2 | 7
Not completed — Early disease progression | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 5
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Number of patients registered to the trial.
Groups:
- Dose Escalation Phase Dose 1.: Crizotinib 250mg OD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day1, then Day 1-21 every 28 day cycle
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  PD-0325901: PD-0325901 2mg - 8mg BD with Run in Day -7 to Day-1 on Cycle 1 Day1, then Day 1-21 every 28 day cycle.
- Dose Escalation Phase Dose 2.: Crizotinib 200mg BD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day1, then Day 1-21 every 28 day cycle
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  PD-0325901: PD-0325901 2mg - 8mg BD with Run in Day -7 to Day-1 on Cycle 1 Day1, then Day 1-21 every 28 day cycle.
- Dose Escalation Phase Dose 3.: Crizotinib 200mg BD Days 1-28 continuously PD-0325901 4mg BD Run in Day -7 to Cycle 1 Day 1, then Day 1-21 every 28 day cycle
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  PD-0325901: PD-0325901 2mg - 8mg BD with Run in Day -7 to Day-1 on Cycle 1 Day1, then Day 1-21 every 28 day cycle.
- Dose Escalation Phase Dose 4.: Crizotinib 200mg BD Days 1-28 continuously PD-0325901 8mg BD Run in Day -7 to Cycle 1 Day1, then Day 1-21 every 28 day cycle
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  PD-0325901: PD-0325901 2mg - 8mg BD with Run in Day -7 to Day-1 on Cycle 1 Day1, then Day 1-21 every 28 day cycle.
- Dose Escalation Phase 5.: Binimetinib 30mg BD continuous administration or Days 1-21 every 28 days. PF-02341066 200mg BD continuous administration
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  PD-0325901: PD-0325901 2mg - 8mg BD with Run in Day -7 to Day-1 on Cycle 1 Day1, then Day 1-21 every 28 day cycle.
  Binimetinib: Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
- Dose Escalation Phase Dose 5a: Binimetinib 30mg BD interval dose administration Days 1-21 every 28 days. PF-02341066 250mg OD continuous administration
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  Binimetinib: Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
- Dose Escalation Phase Dose 5 (Interval Dosing): Binimetinib 30mg BD interval dose administration days 1-21 every 28 days. PF-02341066 200mg BD continuous administration
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  Binimetinib: Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
- Total: Total of all reporting groups
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4. | Dose Escalation Phase 5. | Dose Escalation Phase Dose 5a | Dose Expansion Phase | Dose Escalation Phase Dose 5 (Interval Dosing) | Total
Number analyzed (Participants) | 6 | 5 | 6 | 8 | 8 | 7 | 37 | 5 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 5 | 5 | 6 | 5 | 24 | 4 | 56
  >=65 years | 2 | 2 | 1 | 3 | 2 | 2 | 13 | 1 | 26
Age, Continuous [Median (Full Range); unit: years] | 65.8 [36 to 78] | 64.8 [48 to 69] | 58.4 [52 to 71] | 61.2 [36 to 73] | 51.0 [33 to 72] | 60.0 [46 to 70] | 62.0 [32 to 78] | 55.0 [40 to 65] | 60.4 [32 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 2 | 3 | 0 | 18 | 3 | 36
  Male | 2 | 2 | 3 | 6 | 5 | 7 | 19 | 2 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Maximal Tolerated Dose (MTD) of PD-0325901 and PF-02341066 /PF-02341066 or Binimetinib With PF-02341066
Description: Determine maximum tolerated dose (MTD) of PD-0325901 with Crizotinib (PF-02341066) according to toxicities graded by NCI CTCAE v4.03, in patients with advanced solid tumours.
Time Frame: Dose Escalation Phase: treatment Cycle 1 28 days (plus 7 day run-in for PD-0325901/PF-02341066 combination)
Population: Evaluable patients are those patients who completed cycle 1 or withdrew early for experiencing a DLT. Four patients withdrew early from the study not for DLTs, consequently 21 patients remained for the dose escalation primary analysis.
Measure: Number; unit: Dose Limiting Toxicities (DLTs)
Groups:
- Dose Escalation Phase Cohort 1 Dose Level 1: Crizotinib (PF-02341066) 250mg OD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day -1, then Day 1-21 every 28 day cycle
- Dose Escalation Phase Cohort 2 Dose Level 2: Crizotinib (PF-02341066) 200mg BD Days 1-28 continuously PD-0325901 2mg BD Run in Day -7 to Cycle 1 Day -1, then Day 1-21 every 28 day cycle
- Dose Escalation Phase Cohort 3 Dose Level 3: Crizotinib (PF-02341066) 200mg BD Days 1-28 continuously PD-0325901 4mg BD Run in Day -7 to Cycle 1 Day -1, then Day 1-21 every 28 day cycle
- Dose Escalation Phase Cohort 4 Dose Level 4: Crizotinib (PF-02341066) 200mg BD Days 1-28 continuously PD-0325901 8mg BD Run in Day -7 to Cycle 1 Day -1, then Day 1-21 every 28 day cycle
Arm/Group | Dose Escalation Phase Cohort 1 Dose Level 1 | Dose Escalation Phase Cohort 2 Dose Level 2 | Dose Escalation Phase Cohort 3 Dose Level 3 | Dose Escalation Phase Cohort 4 Dose Level 4
Number analyzed (Participants) | 6 | 5 | 4 | 6
Dose Limiting Toxicities (DLTs) | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Dose Escalation Phase Cohort 1 Dose Level 1 vs Dose Escalation Phase Cohort 2 Dose Level 2 vs Dose Escalation Phase Cohort 3 Dose Level 3 vs Dose Escalation Phase Cohort 4 Dose Level 4; Test type: Other; The primary dose escalation analysis was to find the MTD, which was defined as the dose of PF-02341066 in combination with PD-0325901 at which no more than one out of six patients experience a DLT (dose limiting toxicity). The DLT was based on observed toxicity in cycle 1, and was defined as an almost certainly or probably drug-related adverse event to PF-02341066 and/or PD-0325901. The MTD for the PD 0325901/PF-02341066 combination was 8mg BD(days1-21) and 200mg BD continuously in a 28 day cycle (Dose Level 4)

2. Primary Outcome: Clinical Response to Binimetinib Combined With PF-02341066
Description: To investigate response to treatment with RPII dose of Binimetinib with Crizotinib (PF-02341066), in patients with a) RASMT CRC or b) RASWT/cMET mut amplified CRC or c) RASWT/c-MET over-expressed CRC, as defined by stable, partially or completely responding disease, per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), Neither sufficient shrinkage to qualify for PR nor sufficient increase (>=20%) to qualify for Progressive Disease; Overall Response (OR) = CR + PR + SD
Time Frame: Dose Expansion phase: change from baseline and up to 12 months.
Population: Evaluable patients for the primary outcome are those patients who complete a response assessment after cycle 1 of treatment, or who progress early on treatment. 30 of the 36 recruited patients had a response assessment after cycle 1 or progressed early on treatment, and hence these 30 patients are evaluable for the primary analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 30
Participants
  Stable Disease | 7
  Progressive Disease | 22
  Early death from malignant disease | 1

3. Primary Outcome: Maximal Tolerated Dose (MTD) of Binimetinib and PF-02341066
Description: To determine the maximal tolerated dose (MTD) of Binimetinib with PF-02341066 according to toxicities graded by NCI CTCAE V4.03 in cycle 1 of treatment.
Time Frame: Dose Escalation Phase: treatment Cycle 1 28 days
Population: Evaluable patients are those patients who completed cycle 1 or who withdraw early for experiencing a DLT. Three patients withdrew early from the study not for DLTs, consequently 17 of the 20 recruited patients are evaluable for this analysis.
Measure: Number; unit: Dose Limiting Toxicities (DLTs)
Groups:
- Dose Escalation Phase Cohort 12 Dose Level 5 (Interval Dosing): Binimetinib 30mg BD interval dose administration Days 1-21 every 28 days. PF-02341066 250mg OD continuous administration
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  Binimetinib: Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
- Dose Escalation Phase Cohort 13 Dose Level 5a: Binimetinib 30mg BD interval dose administration days 1-21 every 28 days. PF-02341066 200mg BD continuous administration
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  Binimetinib: Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
Arm/Group | Dose Escalation Phase Cohort 7 Dose Level 5 | Dose Escalation Phase Cohort 12 Dose Level 5 (Interval Dosing) | Dose Escalation Phase Cohort 13 Dose Level 5a
Number analyzed (Participants) | 6 | 5 | 6
Dose Limiting Toxicities (DLTs) | 2 | 2 | 1
Statistical Analysis 1: Comparison: Dose Escalation Phase Cohort 7 Dose Level 5 vs Dose Escalation Phase Cohort 12 Dose Level 5 (Interval Dosing) vs Dose Escalation Phase Cohort 13 Dose Level 5a; The primary dose escalation analysis was to find the MTD, which was defined as the dose of PF-02341066 in combination with Binimetinib at which no more than one out of six patients experience a DLT (dose limiting toxicity). The DLT was based on observed toxicity in cycle 1, and was defined as an almost certainly or probably drug-related adverse event to PF-02341066 and/or Binimetinib; Test type: Other; Binimetinib 30mg BD on days 1 - 21 every 28 days with Crizotinib 250 mg OD continuously is the MTD, the recommended dose and schedule for further evaluation in our and other trials. This was as only one DLT was experienced in 6 evaluable patients at this final dose escalation level

4. Secondary Outcome: Pharmacokinetic Peak Plasma Concentration (Cmax) for PF-02341066 and PD-0325901.
Description: To investigate the pharmacokinetics (PK) plasma Cmax of PD-0325901 (and its metabolite, PD-0315209) with PF-023241066 when administered in combination.
Time Frame: Dose Escalation:Up to 12 months. PK profile at pre-dose and up to 10 hrs post dose on Day - 1, Day 21 and Day 28 of Cycle 1
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4.
Number analyzed (Participants) | 6 | 4 | 3 | 4
ng/ml
  Summary PD-0325901 PK Day -1 | 77.8 (41.9) | 129 (50.5) | 226 (66.1) | 484 (84.1)
  Summary PD-0325901 PK Day 21 | 70.3 (43.1) | 62.3 (34.7) | 135 (36.2) | 219 (93.6)
  Summary PD-0315209 PK Day -1 | 53.1 (30.7) | 59.4 (35.3) | 117 (44.3) | 195 (55.6)
  Summary PD-0315209 PK Day 21 | 52.0 (24.8) | 46.7 (29.5) | 103 (40.5) | 117 (57.6)
  Summary PF-02341066 PK Day 21 | 170 (81.3) | 300 (53.9) | 235 (35.3) | 269 (157)
  Summary PF-02341066 PK Day 28 | 164 (59.8) | 281 (118) | 341 (133) | 275 (105)

5. Secondary Outcome: Pharmacokinetic Minimum Plasma Trough Concentration (Cmin) for PF-02341066 and PD-0325901
Description: To investigate the pharmacokinetics (PK) plasma Cmin of PD-0325901 (and its metabolite, PD-0315209) with PF-023241066 when administered in combination.
Time Frame: Dose Escalation:Up to 12 mths. Cycle 1 PK profile up to 10 hrs post dose on Day -1, 21 and 28
Population: PK analysis performed on Cycle 1 Day -1 and Day 21 only for PD-0325901 and PD-0315209 and on Cycle 1 Day 21 and Day 28 only for PF-02341066 according to dosing schedule Day -7 to Day 21 for PD-0325901 and Day 1 to Day 28 for PF-02341066.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4.
Number analyzed (Participants) | 6 | 4 | 3 | 4
ng/ml
  Summary PD-0325901 PK Day -1 | 23.6 (9.3) | 18.7 (5.83) | 37.9 (5.89) | 89.2 (24.3)
  Summary PD-0325901 PK Day 21 | 26.0 (16.1) | 17.6 (3.12) | 35.8 (13.3) | 45.4 (13.0)
  Summary PD-0315209 PK Day -1 | 44.0 (29.6) | 40.4 (26.3) | 80.6 (22.1) | 147 (47.7)
  Summary PD-0315209 PK Day 21 | 41.3 (23.3) | 37.3 (25.4) | 66.6 (18.8) | 73.1 (31.7)
  Summary PF-02341066 PK Day 21 | 115 (64.4) | 186 (55.8) | 172 (43.6) | 203 (121)
  Summary PF-02341066 PK Day 28 | 119 (44.4) | 183 (66.3) | 259 (96.0) | 211 (78.6)

6. Secondary Outcome: Pharmacokinetic Area Under the Plasma Concentration Versus Time Curve (AUC) for PF-02341066 and PD-0325901(and Its Metabolite)
Description: To investigate the pharmacokinetics (PK) plasma AUC of PD-0325901 (and its metabolite, PD-0315209) with PF-023241066 when administered in combination.
Time Frame: Dose Escalation:Up to12 months. Cycle 1 PK profile up to 10 hrs on Day -1, 21 and 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4.
Number analyzed (Participants) | 6 | 4 | 3 | 4
ng*hr/mL
  Summary PD-0325901 PK Day -1 | 400 (117) | 432 (129) | 796 (120) | 1907 (254)
  Summary PD-0325901 PK Day 21 | 400 (160) | 301 (106) | 683 (51.7) | 1162 (190)
  Summary PD-0315209 PK Day -1 | 498 (304) | 508 (318) | 954 (301) | 1726 (501)
  Summary PD-0315209 PK Day 21 | 487 (226) | 413 (273) | 831 (246) | 1092 (228)
  Summary PF-02341066 PK Day 21 | 1341 (688) | 2115 (448) | 2034 (397) | 2336 (1414)
  Summary PF-02341066 PK Day 28 | 1378 (567) | 2358 (905) | 2919 (1207) | 2402 (873)

7. Secondary Outcome: Pharmacokinetic Plasma Oral Clearance for PF-02341066 and PD-0325901
Description: To investigate the pharmacokinetics (PK) plasma oral clearance of PD-0325901 (and its metabolite, PD-0315209) with PF-023241066 when administered in combination.
Time Frame: Dose Escalation:Up to12 months.PK profile at Cycle 1 up to 10 hrs post dose on Days -1, 21 and 28
Population: Oral clearance could not be calculated, as pre-specified, as bioavailability and full Area Under the Curve (AUC) data, specifically 0 to ∞ (infinity), was not available. Even though AUC data is available on Days -1, 21 and 28 for 0-10 hours, residual drug at time of next twice daily dose administration meant oral clearance could not be determined for most patients.
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4.
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Progression Free Survival (Dose Expansion)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a >=20% increase in the sum of diameters of target lesions (also demonstrating an absolute increase of at least 5mm) or the appearance of new lesions.
Time Frame: From date of study entry until the date of progression or date of death, assessed up to study completion, an average of 6 months (dose expansion)).
Population: All 37 registered patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Expansion Phase: All of the patients registered for this expansion phase are included in this survival analysis, to preliminarily assess the efficacy of the drug combination.
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 37
months | 1.81 [1.51 to 1.91]

9. Secondary Outcome: Overall Survival (Dose Expansion)
Description: Overall survival (dose expansion).
Time Frame: From date of study entry until the date of death, assessed up to study completion, an average of 6 months (dose escalation).
Population: All 37 registered patients are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 37
months | 5.42 [2.79 to 7.33]

10. Secondary Outcome: Pharmacokinetic (PK) Peak Plasma Concentration (Cmax) for PF-02341066 and Binimetinib.
Description: To investigate the pharmacokinetic (PK) peak plasma concentration (Cmax) of PF-02341066 and Binimetinib and its metabolite, AR00426032, in blood.
Time Frame: Dose Expansion: PK profile up to 10 hrs at Cycle 1 Day 21
Population: Data not available for 2 patients in PF-02341066 outcome measure and 8 patients each in binimetinib and AR00426032 outcome measures
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 26
ng/ml
  Summary PF-02341066 PK Cycle 1 D21 up to 10h: number analyzed (Participants) | 24
  Summary PF-02341066 PK Cycle 1 D21 up to 10h | 197 (112)
  Summary binimetinib PK Cycle 1 D21 up to 10h: number analyzed (Participants) | 18
  Summary binimetinib PK Cycle 1 D21 up to 10h | 357 (171)
  Summary AR00426032 PK Cycle 1 D21: number analyzed (Participants) | 18
  Summary AR00426032 PK Cycle 1 D21 | 22.7 (16.0)

11. Secondary Outcome: Pharmacokinetic Minimum Plasma Trough Concentration (Cmin) for PF-02341066 and Binimetinib.
Description: To investigate pharmacokinetic plasma trough concentration Cmin of PF-02341066 and Binimetinib and its metabolite, AR00426032, in blood.
Time Frame: Dose Expansion: PK profile on Cycle 1 Day 21 up to 10 hrs .
Population: No data available for 8 patients for binimetinib outcome and for 16 patients in AR00426032 outcome measure.
Measure: Mean (Standard Deviation); unit: Cmin (ng/ml)
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 26
Cmin (ng/ml)
  Summary PF-02341066 PK Cycle 1 D21 up to 10h: number analyzed (Participants) | 24
  Summary PF-02341066 PK Cycle 1 D21 up to 10h | 149 (85.3)
  Summary binimetinib PK Cycle 1 D21 up to 10h: number analyzed (Participants) | 18
  Summary binimetinib PK Cycle 1 D21 up to 10h | 103 (58.5)
  Summary AR00426032 PK Cycle 1 D21: number analyzed (Participants) | 18
  Summary AR00426032 PK Cycle 1 D21 | 12.1 (4.80)

12. Secondary Outcome: Pharmacokinetic Area Under the Plasma Concentration Versus Time Curve (AUC) for PF-02341066 and Binimetinib.
Description: To investigate pharmacokinetic area under the plasma concentration versus time curve (AUC) of PF-02341066 and Binimetinib in blood.
Time Frame: Dose Expansion: PK profile on Cycle 1 Day 21 up to 10 hrs
Population: No data available for 2 patients in PF-02341066 outcome measure, 8 for binimetinib outcome measure and 13 for AR00426032 outcome measure
Measure: Mean (Standard Deviation); unit: ng.h/ml (0-10h )
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 26
ng.h/ml (0-10h )
  Summary PF-02341066 PK Cycle 1 D21 up to 10h: number analyzed (Participants) | 24
  Summary PF-02341066 PK Cycle 1 D21 up to 10h | 3478 (2083)
  Summary binimetinib PK Cycle 1 D21 up to 10h: number analyzed (Participants) | 18
  Summary binimetinib PK Cycle 1 D21 up to 10h | 2129 (1152)
  Summary AR00426032 PK Cycle 1 D21: number analyzed (Participants) | 18
  Summary AR00426032 PK Cycle 1 D21 | 194 (85.2)

13. Secondary Outcome: Pharmacokinetic Oral Clearance for PF-02341066 and Binimetinib.
Description: To investigate pharmacokinetic (PK) oral clearance of PF-02341066 and Binimetinib in blood.
Time Frame: Dose Escalation: PK profile at up to 10 hrs post dose on Cycle 1 Day 21
Population: Oral clearance could not be calculated, as pre-specified, as bioavailability and full Area Under the Curve (AUC) data, specifically 0 to ∞ (infinity), was not available. Even though AUC data is available on Day 21 for 0-10 hours, residual drug at time of next twice daily dose administration meant oral clearance could not be determined for most patients.
Arm/Group | Dose Escalation Phase 5. | Dose Escalation Phase Dose 5a | Dose Escalation Phase Dose 5 (Interval Dosing)
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Pharmacodynamic (PD) Effect of PF-02341066 in Combination With PD-0325901 or Binimetinib in Paired Skin Biopsies - Measurement of phosphoMEK1/2.
Description: Measurement of phosphoMEK1/2 in skin biopsies to investigate the pharmacodynamic (PD) effect of PF-02341066 in combination with PD-0325901 or Binimetinib in paired skin biopsies to determine objective response to treatment.
  Western blots are used to measure levels of expression and images are taken of the gels. Image J is used to measure pixels. The minimum is 0 and there is no maximum.
Time Frame: Dose Escalation and Expansion: at baseline and Cycle1, D15.
Population: For the Dose Escalation phases of the study the paired skin biopsies were collected and analysed for eligible patients (achieving end of Cycle 1) where available. Samples for Collection of paired skin biopsies were mandatory for first 10 patients registered to the expansion phase of the study only. An additional 3 samples were collected and analysed in the Expansion phase due to multiple screening performed over several participating sites.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Dose Escalation Phase 5.: Binimetinib 30mg BD continuous administration. PF-02341066 200mg BD continuous administration
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4. | Dose Escalation Phase 5. | Dose Escalation Phase Dose 5a | Dose Escalation Phase Dose 5 (Interval Dosing) | Dose Expansion Phase
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 5 | 5 | 3 | 13
ratio | 3.74 (2.366) | 1.89 (1.425) | 6.52 (5.982) | 5.74 (3.067) | 1.93 (0.844) | 1.03 (0.28) | 0.93 (0.418) | 1.11 (0.697)

15. Secondary Outcome: Pharmacodynamic (PD) Effect of PF-02341066 in Combination With PD-0325901 or Binimetinib in Paired Tumour Biopsies (Where Possible).
Description: Measurement of pSTAT3Y705 to investigate the pharmacodynamic (PD) effect of PF-02341066 in combination with PD-0325901 or Binimetinib in paired tumour biopsies to determine objective response to treatment. Western blots are used to measure levels of expression and images are taken of the gels. Image J is used to measure pixels. The minimum is 0 and there is no maximum.
Time Frame: Dose Escalation: Biopsies at baseline and Cycle1 D15 - both optional.
Population: Biopsies optional for this phase and only consented to by 2 patients for the combination of PF-02341066 with Binimetinib.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Dose Escalation Phase: Binimetinib 30mg BD interval dose administration Days 1-21 every 28 days PF-02341066 (Crizotinib) 250mg OD Days 1-28 continuously Dosage determined following the recommended Phase II dose identification in the dose escalation phase.
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  Binimetinib: Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
Arm/Group | Dose Escalation Phase
Number analyzed (Participants) | 2
ratio | 0.35 (0.2687)

16. Secondary Outcome: Pharmacodynamic (PD) Effect of PF-02341066 in Combination With Binimetinib in Paired Tumour Biopsies (Where Possible).
Description: Measurement of phosphoERK1/2 to investigate the pharmacodynamic (PD) effect of PF-02341066 in combination with Binimetinib in paired tumour biopsies (where possible) to determine objective response to treatment. Western blots are used to measure levels of expression and images are taken of the gels. Image J is used to measure pixels. The minimum is 0 and there is no maximum.
Time Frame: Dose Expansion: Biopsies at baseline and Cycle1 D15. Optional metastic tumour biopsy within 28 days following radiological confirmation of disease progression.
Population: Most patients in expansion phase did not have biopsy collection at Day 15 despite consenting to this procedure prior to commencement of the trial mainly for ethical reasons or inability to access suitable tumour biopsy site.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 2
ratio | 0.155 (0.0212)

17. Secondary Outcome: Progression Free Survival (Dose Escalation Binimetinib/PF-02341066).
Description: as for outcome 8
Time Frame: From date of study entry until the date of progression or date of death, assessed up to study completion, an average of 6 months
Population: All patients registered for this escalation phase are included in this Intention to Treat analysis, as the number of patients in each arm are separately too small for survival analysis, and it is only to preliminarily assess efficacy of the drug. The data is presented as pre-specified in the Statistical Analysis Plan Version 1.0_09Jun2016.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Escalation Phase Binimetinib/PF-02341066: All of the patients registered for this escalation phase are included in this progression free analysis, to preliminarily assess the efficacy of the drug combination.
Arm/Group | Dose Escalation Phase Binimetinib/PF-02341066
Number analyzed (Participants) | 20
months | 2.3 [1.78 to 5.36]

18. Secondary Outcome: Overall Survival (Dose Escalation Binimetinib/PF-02341066)
Description: Overall survival (Dose escalation Binimetinib/PF-02341066).
Time Frame: From date of study entry until the date of death, assessed up to study completion, an average of 6 months
Population: All patients registered for this escalation phase are included in this Intention to Treat analysis, as the number of patients in each arm are separately too small for survival analysis, and it is only to preliminarily assess efficacy of the drug. The data is present as pre-specified in the Statistical Analysis Plan Version 1.0_09June2016.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Dose Escalation Phase Binimetinib/PF-02341066: All of the patients registered for this escalation phase are included in this survival analysis, to preliminarily assess the efficacy of the drug combination.
Arm/Group | Dose Escalation Phase Binimetinib/PF-02341066
Number analyzed (Participants) | 20
months | 8.78 [5.16 to 14.5]

19. Secondary Outcome: Pharmacokinetic Peak Plasma Concentration (Cmax) for PF-02341066 and Binimetinib.
Description: To investigate the pharmacokinetics (PK) plasma Cmax of Binimetinib (and its metabolite AR00426032) with PF-023241066 when administered in combination.
Time Frame: Dose Escalation:Up to 12 months. PK profile at pre-dose and up to 10 hrs post dose on Day 21 of Cycle 1
Population: Dose Escalation phase using binimetinib with PF-02341066. Sample data not available in each outcome measure for 2 patients in Dose level 5 and 1 in Dose level 5 (interval dosing) .
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Dose Escalation Phase Dose 5: Binimetinib 30mg BD continuous administration or Days 1-21 every 28 days. PF-02341066 200mg BD continuous administration
  PF-02341066: PF-02341066 (Crizotinib) 250mg OD or 200mg BD or 250mg BD Days 1-28 continuously
  PD-0325901: PD-0325901 2mg - 8mg BD with Run in Day -7 to Day-1 on Cycle 1 Day1, then Day 1-21 every 28 day cycle.
  Binimetinib: Binimetinib 30mg or 45 mg BD either continuously or Days 1-21 every 28 days
Arm/Group | Dose Escalation Phase Dose 5 | Dose Escalation Phase Dose 5 (Interval Dosing) | Dose Escalation Phase Dose 5a
Number analyzed (Participants) | 5 | 4 | 6
ng/ml
  Summary PF-02341066 PK Cycle 1 D21 up to 10h | 273 (118) | 250 (145) | 186 (36.8)
  Summary binimetinib PK Cycle 1 D21 up to 10h | 265 (83.4) | 386 (189) | 320 (136)
  Summary AR00426032 PK Cycle 1 D21 | 25.1 (15.1) | 29.5 (8.62) | 23.4 (8.04)

20. Secondary Outcome: Pharmacokinetic (PK) Minimum Plasma Trough Concentration (Cmin) for PF-02341066 and Binimetinib.
Description: To investigate the pharmacokinetic (PK) minimum plasma trough concentration (Cmin) of PF-02341066 and binimetinib in blood.
Time Frame: Dose Escalation phase :Up to 12 months. PK profile at pre-dose and up to 10 hrs post dose on Day 21 of Cycle 1
Population: No data available for 4 patients in dose level 5, for 2 patients in dose level 5 (interval dosing) and for 1 patient in dose level 5a
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Dose Escalation Phase Dose 5 | Dose Escalation Phase Dose 5 (Interval Dosing) | Dose Escalation Phase Dose 5a
Number analyzed (Participants) | 3 | 3 | 5
ng/ml
  Summary PF-02341066 PK Cycle 1 D21 up to 10h | 205 (78.0) | 181 (136) | 114 (43.1)
  Summary binimetinib PK Cycle 1 D21 up to 10h | 77.1 (40.3) | 85.8 (51.9) | 64.0 (28.9)
  Summary AR00426032 PK Cycle 1 D21 | 10.4 (2.66) | 10.2 (2.47) | 6.95 (1.60)

21. Secondary Outcome: Pharmacokinetic Area Under the Plasma Concentration Versus Time Curve (AUC) for PF-02341066 and Binimetinib.
Description: To investigate the pharmacokinetic (PK) area under the plasma concentration versus time curve (AUC) of PF-02341066 and Binimetinib in blood.
Time Frame: Dose Escalation :Up to 12 months. PK profile pre-dose and up to 10 hrs post dose on Day 21 of Cycle 1
Population: No data available for dose level 5 for 3 patients and for 2 patients in dose level 5 (interval dosing)
Measure: Mean (Standard Deviation); unit: ng.h/ml (0-10h )
Arm/Group | Dose Escalation Phase Dose 5 | Dose Escalation Phase Dose 5 (Interval Dosing) | Dose Escalation Phase Dose 5a
Number analyzed (Participants) | 4 | 3 | 6
ng.h/ml (0-10h )
  Summary PF-02341066 PK Cycle 1 D21 up to 10h | 2481 (980) | 2119 (1341) | 1467 (410)
  Summary binimetinib PK Cycle 1 D21 up to 10h | 1604 (554) | 1780 (706) | 1402 (666)
  Summary AR00426032 PK Cycle 1 D21 | 203 (112) | 183 (24.8) | 121 (28.9)

22. Secondary Outcome: Pharmacokinetic Plasma Oral Clearance for PF-02341066 and Binimetinib
Description: To investigate the pharmacokinetics (PK) plasma oral clearance of binimetinib (and its metabolite,AR00426032 ) with PF-023241066 when administered in combination.
Time Frame: Dose Expansion phase at Cycle 1 Day 21 up to 10 hours binimetinib and its metabolite, AR00426032, and up to 24 hours for PF-02341066
Population: as for outcome 13
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 0

23. Secondary Outcome: Pharmacodynamic (PD) Effect of PF-02341066 in Combination With PD-0325901 or Binimetinib in Paired Skin Biopsies - Measurement of phosphoERK1/2.
Description: Measurement of phosphoERK1/2 to investigte the pharmacodynamic (PD) effect of PF-02341066 in combination with PD-0325901 or Binimetinib in paired skin biopsies to determine objective response to treatment. Western blots are used to measure levels of expression and images are taken of the gels. Image J is used to measure pixels. The minimum is 0 and there is no maximum.
Time Frame: Dose Escalation and Expansion: at baseline and Cycle1, D15.
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4. | Dose Escalation Phase 5. | Dose Escalation Phase Dose 5a | Dose Escalation Phase Dose 5 (Interval Dosing) | Dose Expansion Phase
Number analyzed (Participants) | 6 | 5 | 5 | 5 | 5 | 5 | 3 | 13
ratio | 0.47 (0.277) | 0.35 (0.356) | 0.49 (0.727) | 0.34 (0.218) | 0.38 (0.238) | 0.69 (0.147) | 0.23 (0.166) | 0.44 (0.309)

24. Secondary Outcome: Pharmacokinetic Plasma t1/2 Etc for PF-02341066 and PD-0325901
Description: To investigate the pharmacokinetics (PK) plasma half life of PD-0325901 (and its metabolite, PD-0315209) with PF-023241066 when administered in combination.
Time Frame: Dose Escalation:Up to12 months.PK profile at Cycle 1 up to 10 hrs post dose on Days -1, 21 and 28
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Dose Escalation Phase Dose 1. | Dose Escalation Phase Dose 2. | Dose Escalation Phase Dose 3. | Dose Escalation Phase Dose 4.
Number analyzed (Participants) | 6 | 4 | 3 | 4
h
  Summary Half Life of PD-0325901 PK Day -1 | 7.9 (4.1) | 16.8 (13.9) | 9.9 (3.2) | 15.1 (12.5)
  Summary Half Life of PD-0325901 PK Day 21 | 4.5 (0.7) | 9.7 (2.8) | 6.3 (3.2) | 24.8 (27.9)
  Summary Half Life of PD-0315209 PK Day -1 | 18.0 (5.66) | 11.3 (1.2) | 16.0 (6.2) | 15.0 (2.0)
  Summary Half Life of PD-0315209 PK Day 21 | 10.6 (4.88) | 19.3 (3.8) | 11.0 (1.4) | 6.6 (0.6)
  Summary Half Life of PF-02341066 PK Day 21 | 31.5 (22.4) | 10.0 (3.0) | 20.0 (12.3) | 16.0 (10.0)
  Summary Half Life of PF-02341066 PK Day 28 | 31.2 (16.3) | 12.0 (3.3) | 18.5 (12.0) | 22.0 (13.4)

25. Secondary Outcome: Pharmacokinetic Plasma t1/2 for PF-02341066 and Binimetinib.
Description: To investigate pharmacokinetic (PK) t1/2 of PF-02341066 and Binimetinib in blood.
Time Frame: Dose Escalation: PK profile at up to 10 hrs post dose on Cycle 1 Day 21
Population: No data available for Half Life for Dose Escalation phase outcome measure for PF-02341066 due to limitations of limited time-points available and missing samples, minimal clearance over the 10hr.
  No data available for 3 patients in dose level 5 and 2 in dose level 5 (interval dosing) and 1 in dose level 5a.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Dose Escalation Phase 5. | Dose Escalation Phase Dose 5 (Interval Dosing) | Dose Escalation Phase Dose 5a
Number analyzed (Participants) | 4 | 3 | 5
h
  Summary Half Life for Binimetinib for PK Day 21 up to 10h | 4.3 (1.7) | 5.5 (2.9) | 4.7 (1.0)
  Summary Half Life for AR00426032 (binimetinib metabolite) for PK Day 21 up to 10h | 4.3 (1.9) | 5.3 (2.2) | 5.4 (1.8)

26. Secondary Outcome: Pharmacokinetic Plasma t1/2 Etc for PF-02341066 and Binimetinib
Description: To investigate the pharmacokinetics (PK) plasma half life of binimetinib (and its metabolite,AR00426032 ) with PF-023241066 when administered in combination.
Time Frame: as for outcome 22
Population: Data not available for 8 patients in PF-02341066 outcome measure, 11 patients in binimetinib outcome measure and 16 patients in AR00426032 outcome measure.
  Data for PF-02341066 taken at 24 hour time point due to once daily dosing.
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Dose Expansion Phase
Number analyzed (Participants) | 26
h
  Summary t1/2 life for PF-02341066 PK Cycle 1 D21 up to 24 h | 21 (11)
  Summary t1/2 life for binimetinib PK Cycle 1 D21 up to 10h | 6.32 (8.06)
  Summary t1/2 life for AR00426032 PK Cycle 1 D21 up to 10 hr | 4.70 (1.39)

ADVERSE EVENTS:
Time Frame: Adverse event monitoring starts from the time the time of consent until study completion, an average of 6 months.
Description: The Investigator will monitor each patient for clinical and laboratory evidence of adverse events on a routine basis throughout the study.
  The numbers for this outcome are presented by phase of study rather than dose level for a comparative review across both escalation and expansion phases as Adverse Events numbers at each dose level are very low, especially when separated by AE term. These events were collected irrespective of dose levels and cannot be separated into individual dose levels.
Groups:
- Dose Escalation Phase 1 PF-02341066 and PD-0325901: Dose Escalation Phase 1 - Crizotinib and PD-0325901
- Dose Escalation Phase 2 PF-0341066 and Binimetinib: Dose Escalation Phase 2 - Binimetinib and PF-02341066
Arm/Group | Dose Escalation Phase 1 PF-02341066 and PD-0325901 | Dose Escalation Phase 2 PF-0341066 and Binimetinib | Dose Expansion Phase
All-Cause Mortality (participants affected / at risk) | 18/25 | 15/20 | 27/36
Serious Adverse Events (participants affected / at risk) | 9/25 | 12/20 | 18/36
Other Adverse Events (participants affected / at risk) | 25/25 | 20/20 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase 1 PF-02341066 and PD-0325901 (N=25) | Dose Escalation Phase 2 PF-0341066 and Binimetinib (N=20) | Dose Expansion Phase (N=36)
Abdominal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ascitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Bowel Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Brain Metastases (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1)
Caridac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Central Serous Retinopathy (Bilateral) (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Colonic Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Cytolysis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Edema Face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Ejection Fraction Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lower Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lung Infection (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Mucositis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Postural hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Postoperative Hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Thromboembolic Event (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Tingling In Lower Limbs (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Worsening Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Escalation Phase 1 PF-02341066 and PD-0325901 (N=25) | Dose Escalation Phase 2 PF-0341066 and Binimetinib (N=20) | Dose Expansion Phase (N=36)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 1 (3) | 5 (7)
Abdominal Pain Lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 3 (5) | 3 (4) | 8 (17)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 7 (9) | 1 (1) | 9 (16)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (5) | 3 (4)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (6) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 3 (4) | 3 (5) | 9 (13)
Asthenia (General disorders) | 2 (2) | 6 (10) | 9 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (4)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Blood Albumin Decreased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood Alkaline Phosphatase Increased (Investigations) | 5 (7) | 0 (0) | 6 (9)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 7 (19) | 11 (25)
Blood Creatinine Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Lactate Dehydrogenase Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Blood Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood Potassium Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Sodium Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Body Temperature Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
C-Reactive Protein Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Candida Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract Operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Chills (General disorders) | 2 (2) | 1 (1) | 0 (0)
Chorioretinopathy (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Cognitive Disorder Cognitive Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (20) | 4 (5) | 9 (12)
Corneal Opacity (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 6 (9) | 1 (4)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 10 (15) | 14 (28) | 18 (29)
Dizziness (Nervous system disorders) | 1 (1) | 4 (5) | 2 (3)
Dizziness Postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (3)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 5 (8)
Ear Disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Edema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema extremities (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema Face (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema Limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema Lower Limb (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema of legs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Ejection Fraction Decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Electrocardiogram Qtc Interval Prolonged (Investigations) | 1 (2) | 0 (0) | 0 (0)
Epigastric Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Exertional Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Expressive Dysphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eyelid Function Disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Facial rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 10 (18) | 10 (16) | 14 (30)
Fever (General disorders) | 2 (2) | 1 (1) | 4 (5)
Finger cramps (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Foot Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Furunculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gamma-Glutamyltransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal Reflux (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Genital Itching Nos (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ggt Increased (Investigations) | 1 (1) | 0 (0) | 2 (2)
Glucose Increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hand Swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 1 (1)
Heartburn (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic Haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Herpes Lesion Intra-Oral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Hot Flushes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (10) | 3 (4) | 3 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypokalaemia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (2) | 0 (0) | 1 (1)
Intercostal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal Stoma Complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Intra-Abdominal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Itchy Scalp (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint Instability (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
K+ Decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Ldh Increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Left Ventricular Ejection Fraction Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Leg Oedema (General disorders) | 2 (2) | 2 (3) | 0 (0)
Libido Decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Liver Pain (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1)
Localised Numbness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Loose Stools (Gastrointestinal disorders) | 1 (3) | 0 (0) | 0 (0)
Low Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Low Mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (3)
Lymphoedema (Vascular disorders) | 1 (5) | 0 (0) | 0 (0)
Macular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Mucositis (General disorders) | 2 (2) | 1 (1) | 1 (2)
Muscle Ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Myalgia Of Lower Extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 11 (20) | 11 (16) | 20 (29)
Nausea And Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathic Pain (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3)
Nose Bleeds (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (4) | 2 (4) | 1 (1)
Oedema Abdomen (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema Arms (General disorders) | 1 (2) | 0 (0) | 0 (0)
Oedema Extremities (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema Legs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema Limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema Of Lower Extremities (General disorders) | 1 (1) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral Candida (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Orofacial Oedema (General disorders) | 1 (1) | 0 (0) | 1 (1)
Osteoarticular Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis Of Jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain In Hip (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Pain In Thigh (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain Jaw (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Painful Hips (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Papular Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 2 (3) | 1 (1) | 0 (0)
Paraesthesia Lower Limb (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Parotiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Periorbital Infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Periorbital Oedema (Eye disorders) | 0 (0) | 3 (3) | 1 (1)
Peripheral Oedema (General disorders) | 0 (0) | 2 (4) | 0 (0)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (2)
Platelet Count Decreased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postprandial Emesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Postural Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Prolapse Of Intestinal Stoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Protein Total Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (6)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pustular Rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Qt Prolonged (Investigations) | 4 (4) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (12) | 11 (21)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 9 (12) | 8 (12) | 13 (19)
Rash Face (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Rash On Legs & Arms (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal Impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Retinal Hemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retrosternal Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rib Pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Right Upper Quadrant Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rigors (General disorders) | 0 (0) | 1 (1) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Runny Nose (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Serous Discharge (General disorders) | 1 (1) | 0 (0) | 0 (0)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2)
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin Peeling (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 0 (0)
Skin Toxicity (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Sodium Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Sore Gums (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Stoma Site Bleeding (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Stomach Cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Subconjunctival Haemorrhage (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Swelling Of Hands (General disorders) | 0 (0) | 1 (1) | 0 (0)
Swelling Of Legs (General disorders) | 1 (1) | 1 (1) | 0 (0)
Teeth Chattering (General disorders) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 1 (4) | 0 (0)
Transaminitis (Investigations) | 0 (0) | 0 (0) | 1
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Urinary Frequency (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (3)
Urine Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vasovagal Attack (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Vision Abnormal (Eye disorders) | 0 (0) | 1 (2) | 0 (0)
Visual Disturbance (Eye disorders) | 3 (3) | 0 (0) | 0 (0)
Visual Field Defect (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (20) | 6 (9) | 19 (37)
Weakness Left Or Right Side (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Weight Gain (Investigations) | 0 (0) | 1 (2) | 0 (0)
Weight Loss (Investigations) | 0 (0) | 0 (0) | 1 (1)
Wheeze (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Wound Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Few patients stayed on treatment beyond cycle 2 so long term tolerability has not been evaluated in depth.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT02510001/Prot_003.pdf
  • Statistical Analysis Plan (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02510001/SAP_001.pdf
  • Informed Consent Form (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/01/NCT02510001/ICF_002.pdf